CLINICAL TRIAL: NCT05005195
Title: Yorkshire Kidney Screening Trial (YKST): a Feasibility Study of Adding Non-contrast Abdominal CT Scan to Chest CT Scan Undertaken in the YLST Randomised Controlled Trial of Community-based CT Screening for Lung Cancer in an at Risk Population to Screen for RCC and Other Abdominal Malignancies
Brief Title: Yorkshire Kidney Screening Trial
Acronym: YKST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Collaborators: University of Cambridge (Other); Yorkshire Cancer Research (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Professor Grant Stewart, Principal Investigator, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 290336
Record Dates: First submitted 2021-08-04; First posted 2021-08-13 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Screening; Feasibility study
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: A non-randomised feasibility study of adding non-contrast CT scanning of the abdomen to the CT chest undertaken in the T2 round of YLST.
  YLST is a two-arm, (1:1) implementation study using a single-consent Zelen's randomised controlled design. Participants have already been randomised to intervention (invitation to an initial telephone-based riskassessment and then, if eligible, for a Lung Health Check (LHC) which is carried out on a mobile van and incorporates LDCT scanning for lung cancer) or usual care (no invitation).
Masking Description: There is no randomisation in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal CT Scan (Other): A policy of invitation to a targeted community-based non-contrast CT screening of the abdomen in those at risk of kidney cancer.
  Interventions: Radiation: Low dose abdominal computed tomography scan

INTERVENTIONS:
Radiation: Low dose abdominal computed tomography scan — A policy of invitation to a targeted community-based non-contrast CT screening of the abdomen in those at risk of kidney cancer

SUMMARY:
Kidney cancer is the 8th most common cancer in Yorkshire. It has a poor survival rate, with only 6 out of 10 patients diagnosed with kidney cancer still alive after 5 years. This is partly because many people with kidney cancer don't have any symptoms. In some of these people, kidney cancer is only found by chance during investigations for other reasons. In others, it is often not diagnosed until the disease has passed the point at which we can easily cure it.

Screening for kidney cancer has the potential to pick up these cancers earlier and increase the number of people who can be cured. The Yorkshire Lung Screening Trial offers people aged 55-80 with a history of smoking a CT scan as part of a lung health check. This group of people is also at increased risk of developing kidney cancer. Our new study, the Yorkshire Kidney Screening Trial, will piggyback on this trial to offer an extra CT scan for kidney cancer. The extra scan will take 10 seconds. By the end of the study we will understand whether it is workable to roll this out more widely and whether people take up this extra scan.

DETAILED DESCRIPTION:
Background to YLST and link with YKST

YKST will be offered to participants of YLST. In brief, YLST is a community-based screening programme funded by Yorkshire Cancer Research which uses mobile units across Leeds through a Zelen's design study, allowing assessment of the overall effect of screening Yorkshire people who are current smokers or ex-smokers and therefore at high-risk for lung cancer. YLST is one of the World's largest lung cancer screening trials and nesting YKST within this on-going trial provides a unique opportunity to both add value to this existing trial and provide much needed data relating to future RCC screening.

In YLST, ~45,000 people were invited to participate in the study with 6,892 eventual participants estimated to attend for the first of two rounds of low-dose CT (LDCT) screening (called T0 and T2 respectively). To identify eligible individuals, General Practices within the Leeds CCG area provided consent for interrogation of their Primary Care databases

At the first Lung Health Check (T0) relevant clinical and demographic information were collected and participants were offered a LDCT scan either immediately or to return another day at their preference. Two years later the participants who attended for an initial Lung Health Check are invited back for a follow-up Lung Health Check (T2) which includes a second LDCT scan. In YKST we are asking participants in this T2 round of YLST, from 10 May 2021 to 31 Oct 2022, to undergo an abdominal CT scan in addition to the repeated CT chest.

Participant pathway and detailed logistics

There are 2 major elements to the logistics of YKST: 1) Obtaining the abdominal CT scan. From invitation to completion of the CT scan, the existing YLST infrastructure will be used on the YLST van. 2) Downstream processes from the scan. Reporting of the CT scan, informing participants of results and dealing with anomalies. These are new YKST specific processes, separate to YLST. Invitation YLST participants will receive a telephone call to book a T2 round appointment. Following this they will receive an appointment letter. If the participant is not available after 2 attempted telephone calls, they are sent a pre-booked appointment.

Consent

On arriving on the YLST van the potential participants will watch the YLST T2 introduction video. Following the YLST T2 introduction video the YKST PIS video will play, this will have been mentioned to YLST participants by van staff on arrival . They will then have the YLST consultation in a private consultation room. After completing the YLST components, they will be asked if they wish to participate in YKST. For those wishing to take part, written consent will be taken whilst in the consultation room and a small number of extra RCC specific questions will be.

Those not wishing to take part will also be asked to give their reasons for declining and asked if they consent to be contacted by a University of Cambridge researcher to discuss taking part in a qualitative interview about their reasons for declining.

Those wishing to have the additional scan will also be asked if they consent to be contacted by a University of Cambridge researcher to discuss taking part in a qualitative research interview about reasons for agreeing to participate. Participants consenting to be contacted by the research team about an interview (those wishing to have the additional scan and those declining the scan) will be sent a separate PIS and a consent form and asked to contact the team if they would like to take part. A member of the research team will then contact them to arrange a convenient time for a telephone or remote video interview. Those taking part will be asked to sign the consent form and send this back to the research team in a stamped addressed envelope, or sign it electronically. In case there is a delay in this process, possibly due to the COVID19 pandemic, verbal consent will also be taken over the telephone at the start of the interview.

All healthcare professionals involved in the screening process will also be invited by the research team to take part in an interview about the acceptability of the combined approach and the logistics. They will be provided with a PIS and consent form and consent taken as for screening participants above.

CT scanning protocol and reporting

Following confirmation that the participant has not has an abdominal CT scan within the previous 6 months, scans will be ordered by the YKST nurse research team or research fellow. We have designed a clear risk mitigation process to ensure that if a participant wishes to continue with lung screening as part of YLST but does not want to participate in the YKST component, that they do not get the abdominal CT scan. The mechanism for this is that a hard copy of the Kidney Screening CT request form will only be printed once participants have signed the YKST consent form. As an additional check the radiographers will be asked to sign the request form to indicate that they have seen the YKST consent form before proceeding to the additional kidney screening scan. This will act as an additional prompt for the radiographer team to ensure that the correct screening protocols are used.

The abdominal CT scan will be performed immediately following the CT chest for YLST, the patient will remain lying the CT scanner gantry and the abdominal CT will take a further 10 seconds to be performed.

Management of screening results

The Lead Consultant Radiologist and the YKST Principal Investigator (a Consultant Urologist)at Leeds Teaching Hospitals NHS Trust have developed a series of pathways for flagging in the CT report, based on: 1 - Normal; 2 - benign urological finding; 3 - Indeterminate benign finding (i.e. cholecystitis/pancreatitis); 4 Possible malignancy outside renal tract (2 week wait referral) or AAA (referral to vascular surgery); 5 - Possible renal/urological cancer (2 week wait referral).

The PI will work with the nurse practitioner and administration support employed by YKST for the duration of the scanning period so that they can inform the patients of results and refer patients to the appropriate other specialities: e.g. vascular and HPB surgery There are no further visits of assessments for participants of YKST.

Qualitative interviews and ethnography

We will conduct semi-structured qualitative telephone or remote video interviews within 3 months of the initial study invitation with a purposive sample of both participants who take up the additional abdominal CT scan and those who decline the additional scan. The interviews will explore their views on the acceptability of the combined screening approach, the consent process, the information provided about the additional scan, and their reasons for accepting or declining the scan. We will also explore potential psychological harms, for example, increased anxiety or worry related to the additional scan or the information provided about kidney cancer and other potential abdominal findings. We will draw on the principles of information power when deciding when to cease data collection but anticipate interviewing up to 40 participants. We will purposefully sample participants with the aim to include approximately 20 who took up the additional scan and 20 who did not and to include participants with a range of ages, sex, and abdominal findings. Interviews will be recorded and transcribed for analysis. We expect interviews to last between 30-45 minutes.

To assess the study processes, including ordering the scans, obtaining consent, ensuring only participants consenting to the additional abdominal scan receive it, performing, reporting and reviewing the additional scans and feeding back the results, from the perspective of the healthcare professionals we will also conduct telephone/video link interviews with key individuals involved in the screening pathway. These will include CTAs, research nurses, radiographers, radiologists and the triaging urologist. The interview schedule will cover their views on all stages of the pathway relevant to them.

To explore in more detail the consent and scanning process on the screening vans, we will also conduct an ethnographic study with a researcher spending time on the vans observing the patient flow and processes. The field notes from these observations will be combined with the analysis of the interview data to enable us to identify aspects that worked well and any challenges or potential safety concerns within the proposed combined screening pathway in order to inform a future RCT.

ELIGIBILITY:
Inclusion criteria

As YKST will involve only consenting participants of T2 round of YLST the same inclusion criteria for the YLST Lung Health Check at the T0 stage will be used for YKST, namely:

High risk for lung cancer as defined by one of the three criteria:

* 30 pack year history of smoking and current smoker or quit within the last 15 years (USPSTF criteria).
* Lung cancer risk of ≥1.51% over 6 years as calculated by the PLCOM2012 score.
* Lung cancer risk of ≥5% over 5 years as calculated by the LLPv2. score.

Exclusion Criteria:

* Have undergone CT Thorax within the previous 6 months
* Unable to provide informed consent to study
* Unable to have a chest or abdominal non-contrast CT scan
* Previous diagnosis of kidney cancer
* Have undergone abdominal CT scan in previous 6 months

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5850 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of individuals who take up the offer of an abdominal CT scan | At the end of the 18 month recruitment period
  The proportion of individuals attending the T2 round of YLST who take up the offer of an abdominal CT scan
The acceptability of the combined lung and RCC screening approach to participants | On completion of the patient interview analysis - by the end of the 18 month recruitment period
  The acceptability to participants of combined lung and RCC screening by non-contrast CT scanning - ascertained by interviews
The acceptability of the combined lung and RCC screening approach to healthcare professionals | On completion of the health care professional interview analysis - by the end of the 18 month recruitment period
  The acceptability to healthcare professionals involved in the screening of combining RCC screening by non-contrast CT scanning with lung cancer screening - ascertained by interviews
The additional time required for the combined screening approach | On completion of the study process observation analysis - by the end of the 18 month recruitment period
  The additional time required for the combined screening approach, including the time to provide information, consent participants, and perform the lengthier CT scan, the time needed by radiologists for reporting the CT scans, and the additional time to review abdominal CT findings

SECONDARY OUTCOMES:
Estimate of the prevalence of RCC | At the end of the 18 month recruitment period
  The proportion of participants found to have an RCC to provide an estimate of the prevalence of RCC found on non-contrast CT screening in 55-80y smokers and ex-smokers
The stage distribution of all RCCs identified, reported as cancer findings with TNM | At the end of the 18 month recruitment period
  The stage distribution of RCC identified through non-contrast CT screening, reported as cancer findings with TNM
The proportion of participants found to have incidental renal findings | At the end of the 18 month recruitment period
  The proportion of participants found to have incidental renal findings (cysts, anatomical variants) on non-contrast CT scanning
The proportion of participants with non-renal findings | At the end of the 18 month recruitment period
  The proportion of participants with non-renal findings i.e. abdominal aortic aneurysms, pancreatic and liver lesions on non-contrast CT scanning
Estimation of the incidence of RCC | At the end of the 18 month recruitment period
  The proportion of RCCs found on the upper pole of participants in T2 who did not have them found in T0 round, to estimate the incidence of RCC over sequential non-contrast CT scans (n.b. lesions in the upper pole of the kidney only)

CONTACTS AND LOCATIONS:
Overall Officials: Grant D Stewart, Principal Investigator — University of Cambridge
Locations (1):
- Leads Teaching Hospitals Trust, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas C, Heathcote L, Sun Y, Callister MEJ, Kitt J, Rossi SH, Shinkins B, Usher-Smith JA, Whyte S, Stewart GD; YKST Study Group. Cost-effectiveness of one-off upper abdominal CT screening as an add-on to lung cancer screening in England. Br J Cancer. 2025 Aug;133(2):239-247. doi: 10.1038/s41416-025-03043-z. Epub 2025 May 14. PMID 40369122
- [Derived] Usher-Smith JA, Godoy A, Burge SW, Burbidge S, Cartledge J, Crosbie PAJ, Eckert C, Farquhar F, Hammond D, Hancock N, Iball GR, Kimuli M, Masson G, Neal RD, Rogerson S, Rossi SH, Sala E, Smith A, Sharp SJ, Simmonds I, Wallace T, Ward M, Callister MEJ, Stewart GD. The Yorkshire Kidney Screening Trial (YKST): protocol for a feasibility study of adding non-contrast abdominal CT scanning to screen for kidney cancer and other abdominal pathology within a trial of community-based CT screening for lung cancer. BMJ Open. 2022 Sep 20;12(9):e063018. doi: 10.1136/bmjopen-2022-063018. PMID 36127097
- See also: YKST twitter account — https://twitter.com/yorkshirekst?lang=en